CLINICAL TRIAL: NCT04712552
Title: In Vivo Measurement of the Accuracy of the "Neurolocate" Module of the Neurosurgical Robot "Neuromate" in Its Application to Deep Brain Stimulation
Acronym: NEUROLOCATE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 19-PP-22
Record Dates: First submitted 2021-01-14; First posted 2021-01-15 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Parkinson Disease; Dystonia; Tremor
MeSH Terms: conditions — Parkinson Disease; Dystonia; Tremor | interventions — Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stereotactic robot-guided deep brain stimulation procedure: Patients requiring a stereotactic robot-guided deep brain stimulation procedure (Parkinson's disease, disabling tremor, dystonia)
  Interventions: Procedure: deep brain stimulation

INTERVENTIONS:
Procedure: deep brain stimulation — On the day of surgery, under general anesthesia, a Fischer ZD frame will be attached to the skull. A T1-weighted 3D MRI with gadolinium will be performed.
  Investigators will plan on this MRI, anatomical targets and deep brain trajectories using the NeuroInspire surgical planning software.
  The patient will be attached to the base of the robot through the frame. Registration will be performed using the Neurolocate method after the acquisition of 3D CT images using the O-arm. The Neurolocate recording is based on radiographic images.The 3D MRI will be merged with the 3D tomography images taken with the O-arm to co-register the trajectories planned on the MRI in the robot space The surgical procedure will be performed as usual by milling the bone at the entry point and inserting under robotic guidance an electrode through a guide tube to the intended target.

SUMMARY:
The purpose of this study is to evaluate the accuracy of the Neurolocate recording system of the neurosurgical robot Neuromate, marketed by Renishaw, in order to optimize surgical procedures, costs and patient comfort.

DETAILED DESCRIPTION:
Robotic neurosurgery has been developed for nearly 25 years and offers neurosurgeons many advantages, including increased precision.

Accuracy is a key point for stereotactic neurosurgical procedures, particularly for deep brain stimulation electrode implantations.

The accuracy of the Neuromate robot was measured in stereotactic framed and frameless mode in vitro and in vivo during stereo-electroencephalography procedures. Investigators also evaluated the actual accuracy of its application in routine deep brain stimulation procedures using a measurement system independent of the robot itself and the manufacturer. We showed that the average in vivo accuracy was 0.86 mm and the maximum error was 1.55 mm. This accuracy is at least similar to the accuracy of stereotactic frame arms and is compatible with the accuracy required in deep brain stimulation procedures.

The Neurolocate device is a new non-invasive, frameless patient matching module designed for use with the Neuromate stereotactic robot.

The main advantages of the Neurolocate system are that it is less invasive than screw-on markers, simplifies the surgical procedure and reduces the duration of the surgery The accuracy of the Neurolocate frameless recording system was evaluated in vitro and in vivo for robotic stereo-electroencephalography trajectories in epileptic patients and compared to the accuracy of conventional recording using a stereotactic frame.

However, the accuracy of the Neurolocate recording system has never been measured in vivo during deep brain stimulation procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 70 years old requiring a stereotactic robot-guided deep brain stimulation procedure
* Signature of the Informed Consent Form
* Affiliation to the French social security system

Exclusion Criteria:

* Contraindication to MRI
* Hypersensitivity to gadoteric acid, meglumine or any product containing gadolinium.
* Anterior and posterior commissure anatomy modifying brain anatomy
* Patient unable to complete the Comfort Questionnaire due to cognitive or speech impairment
* Pregnant or breastfeeding women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring a stereotactic robot-guided deep brain stimulation procedure (Parkinson's disease, disabling tremor, dystonia)
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2023-01-07 (Actual)

PRIMARY OUTCOMES:
Euclidean distance between the point theoretically aimed at by the robot and the point actually reached | Day of intervention
  Precision measurement: Comparison of the Euclidean distance between the point theoretically aimed at by the robot and the point actually reached, based on their respective stereotactic coordinates with respect to the anterior and posterior commissure line

SECONDARY OUTCOMES:
Occupancy time of the operating room | Day of intervention
  Occupancy time of the operating room between the entry of the patient into the operating room and his exit, comparing the methods based on Neurolocate and the classical method with frame (historical data)
comfort of the patient | Within 3 days after intervention
  Evaluation of the invasiveness of the technique and the comfort of the patient through postoperative interviews, assessing their comfort on a 10-point scale and comparing methods based on Neurolocate and the classic "frame-based" method (historical data).

CONTACTS AND LOCATIONS:
Overall Officials: Denys FONTAINE, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Department of neurosurgery, Nice, France

REFERENCES:
- [Derived] Almairac F, Leplus A, Mondot L, Fontaine D. A New Noninvasive Frameless Registration System for Stereotactic Cranial Biopsy: A Technical Note. Oper Neurosurg. 2023 Jan 1;24(1):64-67. doi: 10.1227/ons.0000000000000426. Epub 2022 Sep 26. PMID 36227183